CLINICAL TRIAL: NCT06680609
Title: The Analgesic Efficacy of Nefopam in Patient Undergoing Orthopedics Surgery with Tourniquet: a Double-blind Case-control Trial
Brief Title: The Analgesic Efficacy of Nefopam in Orthopedics Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, anas munir alrusan, Assistant Professor of Anesthesia, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 52/163/2023
Record Dates: First submitted 2024-11-02; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Pain Management; Orthopedic Procedure Pain
Keywords: opioid; nefopam; tourniquet; orthopedic
MeSH Terms: conditions — Agnosia | interventions — Nefopam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nefopam group (Placebo Comparator)
  Interventions: Drug: Nefopam 20 MG/ML
- Placebo (Other)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nefopam 20 MG/ML — The unlabeled interventional drug solution was administered one at the beginning of surgery. A 10 mL solution containing nefopam 20 mg was infused over 20 min
  Arms: Nefopam group
Drug: Placebo — The unlabeled interventional drug solution was administered one at the beginning of surgery. A 10 mL solution containing placebo diluted with normal saline was infused over 20 min
  Arms: Placebo

SUMMARY:
Pain-free and relief are one of the anesthesiologist's most important concerns during the operation. General aim is always to effectively control pain but while simultaneously reducing opioid requirements to reduce opioid related side effects and mortality. Patients undergoing orthopedic operations tend to have high pain scores and analgesic requirements. In this study, the investigators aim to investigate the effect of adding nefopam on reducing the postoperative pain scores and the need for opioids.

This double-blind placebo-controlled prospective study aims to determine the effectiveness of nefopam in relieving the pain resulting from the operation in addition to the pain resulting from tourniquet. The unlabeled drug solution was administered one at the beginning of surgery. A 10 mL solution containing nefopam 20 mg or placebo diluted with normal saline was infused over 20 min. 11-point visual analogue scale was utilized to assess the pain score.

DETAILED DESCRIPTION:
Nefopam is a non-opioid, non-steroidal, centrally acting analgesic drug that is derivative of the non-sedative benzoxazocine, developed and known in 1960s as fenazocine. Although the mechanisms of analgesic action of nefopam are not well understood, they are similar to those of triple neurotransmitter (serotonin, norepinephrine, and dopamine) reuptake inhibitors and anticonvulsants. It has been used mainly as an analgesic drug for nociceptive pain, as well as a treatment for the prevention of postoperative shivering and hiccups. Based on nefopam's mechanisms of analgesic action, it is more suitable for the treatment of neuropathic pain. The recently discovered dual analgesic mechanisms of action, namely, a) descending pain modulation by triple neurotransmitter reuptake inhibition similar to antidepressants, and b) inhibition of long-term potentiation mediated by N-methyl-D-aspartate (NMDA) from the inhibition of calcium influx like gabapentinoid anticonvulsants or blockade of voltage-sensitive sodium channels like carbamazepine, enable nefopam to be used as a therapeutic agent to treat neuropathic pain. The investigators believe that nefopam could be a viable, safe and cost-effective choice to reduce pain scores resulting from orthopedic surgeries in addition to pain resulting from tourniquet insertion and reduce opioid requirements simultaneously with minimal side effects.

This study is a prospective, double-blind, case-control study conducted at the King Abdullah University Hospital in Jordan during the period of June 2023 to December 2023. The study protocol was approved by the Institutional Review Board of King Abdullah University Hospital and registered at the Clinical Research Information Service. Written informed consent was obtained from all participants before enrollment.

Eligible participants for this study included patients undergoing orthopedic surgery which involved usage of tourniquet under general anesthesia. Only patients aged 15-60 were included in the study. The exclusion criteria were as follows: patients with any contraindication to nefopam, surgery with tourniquet time more than 180 min, patients on opioid medications, patients with preexisting chronic pain syndromes, patients refuse to participate in the study and patients with psychiatric diseases. All participants were randomly divided into two groups (control and nefopam) in a 1:1 ratio using computer-generated randomization. A pharmacist who was not involved in this study handled normal saline or nefopam to the anesthesiologist according to the assigned group with the same drug labeling to ensure double blindness.

Intervention and anesthetic protocol Standard monitoring including electrocardiography, non-invasive blood pressure monitor, pulse oximetry, capnography, and neuromuscular monitoring, was applied to the patients throughout the procedure. Induction was performed using propofol 2mg/kg fentanyl 2 μg/kg and atracurium 0.5mg /kg. Inhalational anesthesia using isoflurane 1- minimum alveolar concentration (MAC) with atracurium was performed to maintain general anesthesia. Mechanical ventilation was controlled to maintain the end-tidal carbon dioxide partial pressure at 30-40 mmHg with an inhaled oxygen fraction of 40%-50%. Body temperature was monitored using an esophageal temperature probe and maintained above 35 °C with a forced air warmer. Neostigmine 2.5 mg with atropine 1mg was used to reverse muscle relaxation at the end of surgery.

The unlabeled interventional drug solution was administered one at the beginning of surgery. A 10 mL solution containing nefopam 20 mg or placebo diluted with normal saline was infused over 20 min. At the end of surgery, all patients were given morphine 0.1 mg/kg or tramadol 1mg/kg for postoperative pain control. Morphine (5 mg) was provided as a rescue analgesic upon the patient's request when the postoperative pain score exceeded 4.

Clinical assessments and outcomes The primary outcome was to compare the severity of pain at the site of surgery and at the site of tourniquet insertion by the use of an 11-point visual analogue scale ranging from 0 (no discomfort) to 10 points (most extreme discomfort).

The secondary outcomes were the amount of opioids used intraoperatively and immediately postoperatively by calculating oral morphine equivalent and the sedation score using postoperative Richmond Agitation-Sedation Scores (RASS).

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing orthopedic surgery which involved usage of tourniquet under general anesthesia.
* Only patients aged 15-60 years

Exclusion Criteria:

* patients with any contraindication to nefopam
* surgery with tourniquet time more than 180 min
* patients on opioid medications
* patients with preexisting chronic pain syndromes
* patients refuse to participate in the study
* patients with psychiatric diseases.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-05-05 (Actual)

PRIMARY OUTCOMES:
The analgesic efficacy of nefopam | 6 months
  The primary outcome was to compare the severity of pain at the site of surgery and at the site of tourniquet insertion by the use of an 11-point visual analogue scale ranging from 0 (no discomfort) to 10 points (most extreme discomfort).
Amount of opioids used intraoperatively | 6 months
  The amount of opioids used intraoperatively and immediately postoperatively by calculating oral morphine equivalent

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdullah University Hospital, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No